CLINICAL TRIAL: NCT03066258
Title: A Phase I/IIa (Phase 1/Phase 2a), Open-label, Multiple-cohort, Dose-escalation Study to Evaluate the Safety and Tolerability of Gene Therapy With RGX-314 in Subjects With Neovascular AMD (nAMD)
Brief Title: Safety and Tolerability of RGX-314 (Investigational Product) Gene Therapy for Neovascular AMD Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RGX-314-001
Record Dates: First submitted 2017-02-17; First posted 2017-02-28 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Neovascular Age-related Macular Degeneration; Wet Age-related Macular Degeneration
Keywords: nAMD; wet AMD; gene therapy

STUDY DESIGN:
Intervention Model Description: dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 3E9 GC (genome copies)/eye of RGX-314 (E means the exponential constant)
  Interventions: Genetic: RGX-314
- Cohort 2 (Experimental): 1E10 GC/eye of RGX-314
  Interventions: Genetic: RGX-314
- Cohort 3 (Experimental): 6E10 GC/eye of RGX-314
  Interventions: Genetic: RGX-314
- Cohort 4 (Experimental): 1.6E11 GC/eye of RGX-314
  Interventions: Genetic: RGX-314
- Cohort 5 (Experimental): 2.5E11 GC/eye of RGX-314
  Interventions: Genetic: RGX-314

INTERVENTIONS:
Genetic: RGX-314 — RGX-314 is a recombinant adeno-associated virus (AAV) gene therapy vector carrying a coding sequence for a soluble anti-VEGF protein

SUMMARY:
Excessive vascular endothelial growth factor (VEGF) plays a key part in promoting neovascularization and edema in neovascular (wet) age-related macular degeneration (nAMD). VEGF inhibitors (anti-VEGF), including ranibizumab (LUCENTIS®, Genentech) and aflibercept (EYLEA®, Regeneron), have been shown to be safe and effective for treating nAMD and have demonstrated improvement in vision. However, anti-VEGF therapy is administered frequently via intravitreal injection and can be a significant burden to the patients. RGX-314 is a recombinant adeno-associated virus (AAV) gene therapy vector carrying a coding sequence for a soluble anti-VEGF protein. The long-term, stable delivery of this therapeutic protein following a 1 time gene therapy treatment for nAMD could potentially reduce the treatment burden of currently available therapies while maintaining vision with a favorable benefit:risk profile.

DETAILED DESCRIPTION:
This Phase I/IIa, open-label, multiple-cohort, dose-escalation study was designed to evaluate the safety and tolerability of RGX-314 gene therapy in subjects with previously treated nAMD. Five doses were studied in approximately 42 subjects. Subjects who met the inclusion/exclusion criteria and had an anatomic response to an initial anti-VEGF injection received a single dose of RGX-314 administered by subretinal delivery. RGX-314 uses an AAV8 vector that contains a gene that encodes for a monoclonal antibody fragment which binds to and neutralizes VEGF activity. Safety was the primary focus for the initial 24 weeks after RGX-314 administration (primary study period). Following completion of the primary study period, subjects continued to be assessed until 104 weeks following treatment with RGX-314.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 50 and ≤ 89 years with a diagnosis of subfoveal CNV (Choroidal neovascularization) secondary to AMD in the study eye receiving prior intravitreal anti-VEGF therapy.
2. BCVA (Best Corrected Visual Acuity) between ≤20/63 and ≥20/400 (≤63 and ≥19 Early Treatment Diabetic Retinopathy Study [ETDRS] letters) for the first patient in each cohort followed by BCVA between ≤20/40 and ≥20/400 (≤73 and ≥19 ETDRS letters) for the rest of the cohort.
3. History of need for and response to anti-VEGF therapy.
4. Response to anti-VEGF at trial entry (assessed by SD-OCT (Spectral Domain Optical Coherence Tomography) at week 1)
5. Must be pseudophakic (status post cataract surgery) in the study eye.
6. AST (Aspartate aminotransferase)/ALT (Alanine aminotransferase) < 2.5 × ULN (Upper limit of normal); TB (Total bilirubin) < 1.5 × ULN; PT (Prothrombin time) < 1.5 × ULN; Hb > 10 g/dL (males) and > 9 g/dL (females); Platelets > 100 × 10^3/µL; eGFR (Estimated glomerular filtration rate) > 30 mL/min/1.73 m^2
7. Must be willing and able to provide written, signed informed consent.

Exclusion Criteria:

1. CNV or macular edema in the study eye secondary to any causes other than AMD.
2. Any condition preventing visual acuity improvement in the study eye, eg, fibrosis, atrophy, or retinal epithelial tear in the center of the fovea.
3. Active or history of retinal detachment in the study eye.
4. Advanced glaucoma in the study eye.
5. History of intravitreal therapy in the study eye, such as intravitreal steroid injection or investigational product, other than anti-VEGF therapy, in the 6 months prior to screening.
6. Presence of an implant in the study eye at screening (excluding intraocular lens).
7. Myocardial infarction, cerebrovascular accident, or transient ischemic attacks within the past 6 months.
8. Uncontrolled hypertension (systolic blood pressure [BP] >180 mmHg, diastolic BP >100 mmHg) despite maximal medical treatment.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-11-24 (Actual); Study Completion 2021-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Heier, MD, Principal Investigator — Ophthalmic Consultants of Boston
Locations (8):
- United States (8):
  - Santa Barbara location, Santa Barbara, California
  - Baltimore location, Baltimore, Maryland
  - Boston location, Boston, Massachusetts
  - Reno location, Reno, Nevada
  - Philadelphia location 1, Philadelphia, Pennsylvania
  - Philadelphia location 2, Philadelphia, Pennsylvania
  - Memphis location, Germantown, Tennessee
  - Houston location, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campochiaro PA, Avery R, Brown DM, Heier JS, Ho AC, Huddleston SM, Jaffe GJ, Khanani AM, Pakola S, Pieramici DJ, Wykoff CC, Van Everen S. Gene therapy for neovascular age-related macular degeneration by subretinal delivery of RGX-314: a phase 1/2a dose-escalation study. Lancet. 2024 Apr 20;403(10436):1563-1573. doi: 10.1016/S0140-6736(24)00310-6. Epub 2024 Mar 27. PMID 38554726

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 3E9 GC (genome copies)/eye of RGX-314 (E means exponential constant)
  RGX-314: RGX-314 is a recombinant adeno-associated virus (AAV) gene therapy vector carrying a coding sequence for a soluble anti-VEGF (Vascular endothelial growth factor) protein
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 6 | 6 | 6 | 12 | 12
Completed | 5 | 6 | 6 | 12 | 11
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: 3E9 GC/eye of RGX-314
  RGX-314: RGX-314 is a recombinant adeno-associated virus (AAV) gene therapy vector carrying a coding sequence for a soluble anti-VEGF protein
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 12 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 6 | 6 | 6 | 12 | 12 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 7 | 6 | 22
  Male | 2 | 3 | 4 | 5 | 6 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 6 | 6 | 12 | 11 | 41
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 5 | 6 | 6 | 11 | 12 | 40
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 12 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: Safety (Participants With Ocular and Non-ocular AEs (Adverse Events) and SAEs (Serious Adverse Events))
Description: Participants with ocular and non-ocular AEs and SAEs through 26 weeks (24 weeks following RGX-314 administration)
Time Frame: 26 weeks (24 weeks following RGX-314 administration)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 12
Participants | 6 | 6 | 6 | 12 | 12

2. Secondary Outcome: Safety (Participants With Ocular and Non-ocular AEs and SAEs)
Description: Participants with ocular and non-ocular AEs and SAEs
Time Frame: 106 weeks (104 weeks following RGX-314 administration)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 12
Participants | 6 | 6 | 6 | 12 | 12

3. Secondary Outcome: Change From Baseline in BCVA (Best Corrected Visual Acuity)
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. A higher score represents better vision.
Time Frame: 106 weeks (104 weeks following RGX-314 administration)
Measure: Mean (Full Range); unit: ETDRS letters
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 5 | 6 | 6 | 12 | 11
ETDRS letters | -7.6 [-16 to 6] | 1.2 [-9 to 8] | 14.0 [-3 to 32] | 0.9 [-45 to 17] | -3.8 [-37 to 8]

4. Secondary Outcome: Change From Baseline in CRT (Central Retinal Thickness)
Description: Retinal fluid status of the study eye was evaluated using spectral domain OCT (Optical Coherence Tomography). A decrease in value indicates a decrease in fluid
Time Frame: 106 weeks (104 weeks following RGX-314 administration)
Measure: Mean (Full Range); unit: μm
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 5 | 6 | 6 | 12 | 11
μm | -88.6 [-248.0 to 11.0] | 25.3 [-10.0 to 110.0] | 2.0 [-46.0 to 142.0] | -56.7 [-170.0 to 160.0] | -108.2 [-360.0 to 85.0]

5. Secondary Outcome: Supplemental Injections (Annualized Rate of Supplemental Injections)
Description: The number of supplemental anti-VEGF injections given after RGX-314 was administered. Injections per year which were determined by the number of supplemental injections divided total follow-up in study days which is annualized to a per year rate. Injections were given for signs of worsening disease at a study visit, per the discretion of the investigator.
Time Frame: 106 weeks (104 weeks following RGX-314 administration)
Measure: Mean (Standard Error); unit: supplemental injections per year
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 12
supplemental injections per year | 10.3 (0.86) | 9.3 (1.94) | 2.8 (1.62) | 4.4 (1.25) | 2.0 (1.07)

6. Secondary Outcome: Mean Change From Baseline in Area of CNV (Choroidal Neovascularization)
Description: Area of Choroidal Neovascularization of the study eye was assessed with color fundus photography. Analysis was performed by the central reading center. An increase in value represents an increase in CNV.
Time Frame: 106 weeks (104 weeks following RGX-314 administration)
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 4 | 5 | 5 | 12 | 11
mm^2 | -0.4 (1.62) | 0.0 (1.24) | -1.2 (1.69) | -1.1 (3.58) | -0.6 (3.30)

ADVERSE EVENTS:
Time Frame: Safety was the primary focus for the initial 24 weeks after RGX-314 administration (primary study period). Following completion of the primary study period, subjects continued to be assessed until 104 weeks following treatment with RGX-314 (Week 106). At the end of the study, subjects were invited to participate in a long-term follow-up study (NCT03999801).
Description: Other AEs reported include: RGX-314-emergent Non-serious Ocular Adverse Events Occurring in >5% of Subjects by Preferred Term, Sorted by Frequency in Total Group As-treated Population
  SAE reported include: RGX-314-emergent Serious Adverse Events by System Organ Class and Preferred Term As-treated Population
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 0/12 | 1/12
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 1/6 | 3/12 | 4/12
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 6/6 | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6) | Cohort 3 (N=6) | Cohort 4 (N=12) | Cohort 5 (N=12)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis Ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6) | Cohort 3 (N=6) | Cohort 4 (N=12) | Cohort 5 (N=12)
Conjunctival Haemorrhage (Eye disorders) | 2 (2) | 3 (3) | 4 (4) | 9 (9) | 11 (11)
Intraocular Pressure Increased (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Visual Acuity Reduced/Impairment (Eye disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 1 (1) — Visual Acuity Reduced & Impairment will be presented as a group term including the AE preferred terms (PTs) of "Visual Acuity Reduced" and "Visual Impairment"
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Eye Pain (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Retinal Degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Photopsia (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Conjunctival Hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Vision Blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Retinal pigmentary changes (depigmentation, pigment epitheliopathy & pigmentation) (Eye disorders) | 0 (0) | 3 (3) | 3 (3) | 12 (12) | 11 (11) — Retinal pigmentary changes is a group term including AE preferred terms of 'Retinal Depigmentation', 'Retinal Pigment Epitheliopathy', and 'Retinal Pigmentation'.
Retinal Haemorrhage (Eye disorders) | 4 (4) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Intraocular Inflammation (Eye disorders) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 2 (2) — Intraocular Inflammation is a group term including AE preferred terms of 'Anterior Chamber Cell', 'Anterior Chamber Flare', and 'Anterior Chamber Inflammation'.
Metamorphopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Retinal Thickening (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Dry Age-Related Macular Degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Erythema Of Eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Posterior Capsule Opacification (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vitreous Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT03066258/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT03066258/SAP_001.pdf